CLINICAL TRIAL: NCT00539812
Title: Brief Intervention to Reduce Drinking and Intimate Partner Violence in Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-STU_016315__0111-001; R01AA016315 (NIH)
Record Dates: First submitted 2007-09-24; First posted 2007-10-05 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Intimate Partner Violence; Substance Use
Keywords: Intimate partner violence; alcohol use; substance use
MeSH Terms: conditions — Substance-Related Disorders; Alcohol Drinking | interventions — Standard of Care; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Standard Care only (standard batterer intervention program)
  Interventions: Behavioral: Standard Care
- 2 (Other): Brief alcohol intervention combined with standard care
  Interventions: Behavioral: Brief Alcohol Intervention combined with standard care

INTERVENTIONS:
Behavioral: Standard Care — Standard 40 hour state mandated batterer intervention program
  Arms: 1
Behavioral: Brief Alcohol Intervention combined with standard care — Brief alcohol intervention combined with standard 40 hour state mandated batterer intervention program
  Arms: 2

SUMMARY:
The purpose of this study is to examine whether adding a brief alcohol treatment to standard violence intervention programs for women will result in reduced drinking, reduced partner violence perpetration, and reduced partner violence victimization. We hypothesize that, relative to standard care, women receiving the additional brief alcohol intervention will have better alcohol use and partner violence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hazardous drinking
* Participation in a batterer intervention program

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2007-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Substance use and intimate partner violence | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Stuart, PhD, Principal Investigator — University of Tennessee-Knoxville & Butler Hospital
Locations (1):
- Butler Hospital & University of Tennessee-Knoxville, Providence, Rhode Island, United States